CLINICAL TRIAL: NCT00003479
Title: Phase II Study of Antineoplastons A10 and AS2-1 Infusions in Patients With Ependymoma
Brief Title: Antineoplaston Therapy in Treating Patients With Ependymoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066516; BC-BT-24 (Other: Burzynski Research Institute, Inc.)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Ependymoma
Keywords: Ependymoma; Anaplastic Ependymoma
MeSH Terms: conditions — Ependymoma | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Patients with an ependymoma will receive Antineoplaston therapy (Atengenal + Astugenal).
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for patients with ependymoma provide limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of patients with ependymoma .

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on patients with ependymoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with ependymoma as measured by an objective response to therapy (complete response, partial response) or stable disease.
* To determine the safety and tolerance of Antineoplaston therapy in patients with ependymoma

OVERVIEW: This is a single arm, open-label study in which patients with ependymoma receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity. After 12 months, patients with a complete or partial response or with stable disease may continue treatment.

To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued to this study

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ependymoma that is unlikely to respond to existing therapy and for which no curative therapy exists
* Evidence of residual tumor (>= 5mm) by MRI scan performed within two weeks prior to study entry
* No brain stem tumors

PATIENT CHARACTERISTICS:

Age:

* 6 months and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm3
* Platelet count greater than 50,000/mm3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No renal failure
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No severe heart disease
* No uncontrolled hypertension
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No severe lung disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study
* No serious active infections or fever
* No other serious concurrent disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulating agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy and recovered (6 weeks for nitrosoureas)
* No concurrent antineoplastic agents

Endocrine therapy:

* Concurrent corticosteroids for cerebral edema allowed (must be on stable dose for at least 1 week prior to study)

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* No prior antineoplaston therapy

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 1966-07; Primary Completion 2000-10 (Actual); Study Completion 2000-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nine patients were recruited between July 1996 and October 2000. All study subjects were seen at the Burzynski Clinic in Houston TX.
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 9
Completed | 6
Not Completed | 3
Not completed — Not evaluable | 3

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: Years] | 7.3 [1.6 to 35.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks; Stable Disease (SD), <50% decrease and <25% increase in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least eight weeks; Progressive Disease (PD), >=25% increase in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 6
Participants
  Partial Response | 1
  Stable Disease | 2
  Progressive Disease | 3

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival
Time Frame: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 9
Percentage of Participants
  6 months overall survival | 66.7
  12 months overall survival | 44.4
  24 months overall survival | 33.3
  36 months overall survival | 22.2
  48 months overall survival | 22.2
  60 months overall survival | 11.1

ADVERSE EVENTS:
Time Frame: 4 years, 2 months
Description: Nine patients were recruited between July 1996 and March 2000. All study subjects were seen at the Burzynski Clinic in Houston TX
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 5/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=9)
Hemoglobin (Blood and lymphatic system disorders) | 1 — The Hemoglobin was not related to Antineoplaston therapy.
Central venous catheter infection (Infections and infestations) | 1 — The Central venous catheter infection was not related to Antineoplaston therapy.
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 1 — The Rash: erythema multiforme was possibly related to Antineoplaston therapy.
Pancreatitis (Gastrointestinal disorders) | 1 — The Pancreatitis was not related to Antineoplaston therapy.
Infection (documented clinically): Blood (Infections and infestations) | 1 — The Infection (documented clinically): Blood was not related to Antineoplaston therapy.
Hypokalemia (Investigations) | 1 — The Hypokalemia was possibly related to Antineoplaston therapy.
Confusion (Nervous system disorders) | 1 — The Confusion was possibly related to Antineoplaston therapy.
Seizure (Nervous system disorders) | 1 — The Seizure was not related to Antineoplaston therapy.
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 — The Somnolence/depressed level of consciousness was not related to Antineoplaston therapy.
Pain: Joint (Musculoskeletal and connective tissue disorders) | 1 — The Pain: Joint was possibly related to Antineoplaston therapy.
Pain: Stomach (Gastrointestinal disorders) | 1 — The Pain: Stomach was not related to Antineoplaston therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=9)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 5
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Central venous catheter infection (Infections and infestations) | 3
Non-functional central venous catheter (General disorders) | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4
Fever (General disorders) | 2
Insomnia (General disorders) | 1
Rigors/chills (General disorders) | 1
Weight gain (General disorders) | 1
Pruritus/itching (General disorders) | 1
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Edema/Fluid retention (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Hemorrhage, GU: Bladder (Renal and urinary disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Infection (documented clinically): Bladder (urinary) (Infections and infestations) | 2
Infection (documented clinically): Blood (Infections and infestations) | 1
Infection (documented clinically): Mucosa (Infections and infestations) | 3
Infection (documented clinically): Pharynx (Infections and infestations) | 1
Infection (documented clinically): Sinus (Infections and infestations) | 1
Infection (documented clinically): Soft tissue NOS (Infections and infestations) | 1
Infection (documented clinically): Urinary tract NOS (Infections and infestations) | 1
Middle ear (otitis media) (Infections and infestations) | 1
Skin (Infections and infestations) | 1
Upper airway (Infections and infestations) | 1
Hyperglycemia (Investigations) | 2
Hypernatremia (Investigations) | 3
Hyperuricemia (Investigations) | 1
Hypocalcemia (Investigations) | 1
Hypochloremia (Investigations) | 1
Hypoglycemia (Investigations) | 1
Hypokalemia (Investigations) | 7
Metabolic/Laboratory - Other (Investigations) | 1
Proteinuria (Investigations) | 1
SGOT (Investigations) | 1
SGPT (Investigations) | 3
Apnea (Nervous system disorders) | 1
Ataxia (incoordination) (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Neuropathy: cranial: CN VIII Hearing and balance (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 3
Somnolence/depressed level of consciousness (Nervous system disorders) | 5
Speech impairment (Nervous system disorders) | 2
Syncope (fainting) (Nervous system disorders) | 1
Pain: Dental/teeth/peridontal (Gastrointestinal disorders) | 1
Pain: Head/headache (Nervous system disorders) | 4
Pain: Joint (Musculoskeletal and connective tissue disorders) | 3
Pain: Stomach (Gastrointestinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No